CLINICAL TRIAL: NCT06013319
Title: Effects of Esmolol on Oxygenation Index by Controlling Heart Rate in Patients With Acute Respiratory Distress Syndrome
Brief Title: Effect of Esmolol on Oxygenation Index in Patients With Acute Respiratory Distress Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhiming Jiang (Other)
Responsible Party: Sponsor-Investigator, Zhiming Jiang, Chief Physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QFSKYLLTZH-2023-043
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: esmolol; ARDS; heart rate; oxygenation index
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — esmolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esmolol group (Experimental): Patients with ARDS who require mechanical ventilation after adequate disease assessment and whose heart rate continues to be ≥95 beats/min, but ≤120 beats/min within 24 hours after diagnosis, for at least 10 minutes without changing the dosage of catecholamine, were diagnosed as atrial fibrillation, atrial flutter or sinus tachycardia. The primary treatment is maintained while the esmolol load dose is administered and the maintenance dose is pumped continuously until the patient's heart rate is maintained between 80 and 94 beats per minute.
  Interventions: Drug: Esmolol
- Control group (No Intervention): Patients with ARDS who need mechanical ventilation after adequate condition assessment and whose heart rate continues to be ≥95 beats /min but ≤120 beats /min after optimal hemodynamic treatment within 24 hours after diagnosis were randomly included in the control group. Routine mechanical ventilation, full sedation and analgesia, maintain RASS score 0-2 points; The target tidal volume is 6ml/kg, and the ventilator parameters should be adjusted in time according to the blood gas analysis. Hypotensive patients with sufficient blood volume should be pumped with pressor drugs. Timely sputum suction, airway management, eliminate fever, asthma, pain and other stimulation caused by the heart rate is too fast.

INTERVENTIONS:
Drug: Esmolol — The load dose of esmolol was first injected intravenously: 0.5mg/kg.min, for about 1 minute; then the maintenance dose was pumped intravenously: from 0.05mg/kg/min, and continued after 4 minutes if the efficacy was ideal; if the efficacy was poor, the load dose could be repeated and the maintenance dose increased by 0.05mg/kg/min. The maintenance dose should not exceed 0.3mg/kg/min.
  Other Names: Esmolol hydrochloride injection
  Arms: Esmolol group

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a clinical syndrome caused by intrapulmonary and/or extrapulmonary causes, characterized by intractable hypoxemia. Studies have shown that the sympathetic nervous system is over-activated in patients with acute respiratory distress syndrome. A large retrospective study showed a reduction in mortality in ARDS patients treated with oral β1 blockers before admission, and this beneficial effect of β1 blockers applies to ARDS patients with or without cardiac disease. Esmolol is an ultra-short-acting selective β1 receptor blocker. Previous studies have shown that esmolol can improve oxygenation and reduce the levels of inflammatory cytokines and exudate proteins in bronchoalveolar lavage fluid, thereby alleviating pulmonary injury. According to the literature and our previous clinical observations, we made the following hypothesis: When Estolol is applied to various ARDS patients undergoing mechanical ventilation in ICU, it can control the heart rate by inhibiting β-adrenergic receptor, which can ultimately improve the oxygenation index of patients and shorten the mechanical ventilation time. This project intends to include ARDS patients with optimal hemodynamic treatment for 24 hours, whose heart rate is still ≥95 beats/min after conventional treatment, but ≤120 beats/min. They are randomly divided into control group and Esmolol treatment group to study the effects of esmolol on patients' oxygenation index, mechanical ventilation time, hemodynamics, function of various organs and inflammation level. The aim of this study is to optimize the treatment of ARDS patients.

DETAILED DESCRIPTION:
At present, there are few studies on Esmolol in acute respiratory distress syndrome. However, previous studies have shown that Esmolol can improve oxygenation and reduce the levels of inflammatory cytokines and exudate proteins in bronchoalveolar lavage fluid, thus alleviating pulmonary injury. Considering that a considerable number of ARDS patients in the intensive care unit suffer from sepsis, we conducted this study to explore the application timing of esmolol therapy and whether esmolol can improve the symptoms and prognosis of ARDS patients. Based on the literature and our previous clinical observations, we make the following assumptions: Esmolol is applied to various ARDS patients receiving mechanical ventilation in ICU. By inhibiting the β-adrenergic receptor to control the heart rate, it can ultimately improve the oxygenation index of patients, shorten the mechanical ventilation time, achieve tracheal intubation extraction as soon as possible, and reduce the 28-day mortality. At the same time, esmolol can also improve the function of various organs of patients and reduce the level of inflammatory factors. This project intends to include ARDS patients with optimal hemodynamic treatment for 24 hours, whose heart rate is still ≥95 beats/min after conventional treatment, but ≤120 beats/min. They are randomly divided into control group and Esmolol treatment group to study the effects of esmolol on patients' oxygenation index, mechanical ventilation time, hemodynamics, function of various organs and inflammation level. To optimize the treatment of ARDS patients.

Acute respiratory distress syndrome (ARDS) is a clinical syndrome caused by intrapulmonary and/or extrapulmonary causes, characterized by intractable hypoxemia. ARDS is the most common cause of respiratory failure in severe patients, and also the main factor leading to poor prognosis in severe patients. In recent years, although the research on ARDS has continued to go deeper, clinical treatment still remains in the stage of lung protective ventilation and restricted fluid management, and there is still a lack of specific drug therapy, and the fatality rate is still as high as 40%.

Studies have shown that the sympathetic nervous system is over-activated in patients with acute respiratory distress syndrome. Because 75 to 80 percent of myocardial adrenergic receptors are β1 type, and adrenergic stress is primarily mediated by beta receptors, the heart is a prime target for sympathetic overstimulation. Elevated heart rate is associated with adverse outcomes in patients with severe infection and represents the severity of the disease.Another large retrospective study showed a reduction in mortality in ARDS patients treated with oral β1 blockers before admission, and this beneficial effect of β1 blockers applies to ARDS patients with or without cardiac disease.

Esmolol is an ultra-short-acting selective β1 receptor blocker, which mainly inhibits β1 receptor by competing for catecholamine binding sites in myocaroma, and has the effect of slowing resting and exercise heart rate, lowering blood pressure, and reducing myocardial oxygen consumption. Esmolol is a metabolite coupled with enzyme, so its distribution half-life is very short, intravenous injection begins to take effect 1-2 min, elimination half-life is only 9min, easy to control, high safety, and remarkable effect. There have been numerous studies on esmolol in sepsis. For patients with septic shock, the use of esmolol can reduce heart rate to the target level, but does not increase the incidence of adverse events, and does not reduce microcirculation perfusion, and can improve the hemodynamics and 28-day mortality of patients. In addition, both animal and human experiments have proved that Esmolol can reduce the release of inflammatory factors in sepsis, improve inflammatory response, and protect cardiac and renal function.

At present, there are few studies on Esmolol in acute respiratory distress syndrome. However, previous studies have shown that Esmolol can improve oxygenation and reduce the levels of inflammatory cytokines and exudate proteins in bronchoalveolar lavage fluid, thus alleviating pulmonary injury. Considering that a considerable number of ARDS patients in the intensive care unit suffer from sepsis, we conducted this study to explore the application timing of esmolol therapy and whether esmolol can improve the symptoms and prognosis of ARDS patients. Based on the literature and our previous clinical observations, we make the following assumptions: Esmolol is applied to various ARDS patients receiving mechanical ventilation in ICU. By inhibiting the β-adrenergic receptor to control the heart rate, it can ultimately improve the oxygenation index of patients, shorten the mechanical ventilation time, achieve tracheal intubation extraction as soon as possible, and reduce the 28-day mortality. At the same time, esmolol can also improve the function of various organs of patients and reduce the level of inflammatory factors. This project intends to include ARDS patients with optimal hemodynamic treatment for 24 hours, whose heart rate is still ≥95 beats/min after conventional treatment, but ≤120 beats/min. They are randomly divided into control group and Esmolol treatment group to study the effects of esmolol on patients' oxygenation index, mechanical ventilation time, hemodynamics, function of various organs and inflammation level. To optimize the treatment of ARDS patients.

To evaluate the effect of Esmolol control on heart rate in patients with acute respiratory distress syndrome (ARDS) on oxygenation index. A total of 187 patients aged 18-65 years who met the 2012 Berlin diagnostic criteria for acute respiratory distress syndrome will be included in our study. Hemodynamic optimization was performed within 24 hours after diagnosis. After treatment, the patient's heart rate continued to be ≥95 beats/min but ≤120 beats/min for at least 10 minutes, with or without esmolol pumping. The improvement of oxygenation index in different treatment groups was observed.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the 2012 Berlin diagnostic criteria for acute respiratory distress syndrome;
* Aged between 18-65 years (inclusive);
* 95 times/min ≤ heart rate ≤120 times/min;
* The patient needs to undergo endotracheal intubation mechanical ventilation after condition assessment;
* Obtain the informed consent of the patient or his legal representative.

Exclusion Criteria:

* Bradycardia and second degree or more atrioventricular block;
* Long-term use of beta-blockers;
* Combined with emphysema, asthma and other β-blocker contraindicated diseases;
* Cardiac insufficiency (NYHA grade Ⅲ or Ⅳ);
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Oxygenation index improved or not | From the start of the trial to 12 hours after administering the drug
  To evaluate the effect of Esmolol control on heart rate in patients with acute respiratory distress syndrome (ARDS) on oxygenation index.
Oxygenation index improved or not | From the start of the trial to 24 hours after administering the drug
  To evaluate the effect of Esmolol control on heart rate in patients with acute respiratory distress syndrome (ARDS) on oxygenation index.
Oxygenation index improved or not | From the start of the trial to 48 hours after administering the drug
  To evaluate the effect of Esmolol control on heart rate in patients with acute respiratory distress syndrome (ARDS) on oxygenation index.
Oxygenation index improved or not | From the start of the trial to 72 hours after administering the drug
  To evaluate the effect of Esmolol control on heart rate in patients with acute respiratory distress syndrome (ARDS) on oxygenation index.
Oxygenation index improved or not | From the start of the trial to 120 hours after administering the drug
  To evaluate the effect of Esmolol control on heart rate in patients with acute respiratory distress syndrome (ARDS) on oxygenation index.

SECONDARY OUTCOMES:
the difference of mechanical ventilation duration | from the start of the trial to removal of the endotracheal tube and cessation of mechanical ventilation，up to 28 days
  The duration of mechanical ventilation was compared between the two groups with or without esmolol treatment

CONTACTS AND LOCATIONS:
Overall Officials: zhiming Jiang, doctor, Study Director — Qianfo Mountain Hospital, Shandong Province
Locations (1):
- Department of Intensive Care Medicine, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meyer NJ, Gattinoni L, Calfee CS. Acute respiratory distress syndrome. Lancet. 2021 Aug 14;398(10300):622-637. doi: 10.1016/S0140-6736(21)00439-6. Epub 2021 Jul 1. PMID 34217425
- [Background] van der Jagt M, Miranda DR. Beta-blockers in intensive care medicine: potential benefit in acute brain injury and acute respiratory distress syndrome. Recent Pat Cardiovasc Drug Discov. 2012 Aug;7(2):141-51. doi: 10.2174/157489012801227274. PMID 22642505
- [Background] Morelli A, Donati A, Ertmer C, Rehberg S, Kampmeier T, Orecchioni A, D'Egidio A, Cecchini V, Landoni G, Pietropaoli P, Westphal M, Venditti M, Mebazaa A, Singer M. Microvascular effects of heart rate control with esmolol in patients with septic shock: a pilot study. Crit Care Med. 2013 Sep;41(9):2162-8. doi: 10.1097/CCM.0b013e31828a678d. PMID 23873274
- [Background] Levy B, Fritz C, Piona C, Duarte K, Morelli A, Guerci P, Kimmoun A, Girerd N. Hemodynamic and anti-inflammatory effects of early esmolol use in hyperkinetic septic shock: a pilot study. Crit Care. 2021 Jan 7;25(1):21. doi: 10.1186/s13054-020-03445-w. PMID 33413583